CLINICAL TRIAL: NCT01453530
Title: Street Fitness in Surgical Patients Undergoing General Anesthesia After Reversal of Neuromuscular Rest Blockade With Sugammadex
Brief Title: Street Fitness in Surgical Patients Undergoing General Anesthesia After Reversal of Neuromuscular Blockade
Acronym: SFINX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35385.091.11
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-09

CONDITIONS: Anesthesia Recovery Period
Keywords: Recovery; Street fitness; Sugammadex; Alertness; Ambulatory surgery
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sugammadex (Active Comparator): A single dose of sugammadex 2 mg/kg iv. Dose calculation will be based on the patient's actual body weight. No dose adjustments are allowed
  Interventions: Drug: Sugammadex
- Neostigmine/glycopyrrolate (Active Comparator): A single dose of neostigmine 0.04 mg/kg iv plus glycopyrrolate 0.01 mg/kg iv. Dose calculation will be based on the patient's actual body weight. No dose adjustments are allowed.
  Interventions: Drug: Neostigmine/Glycopyrrolate
- No reversal agent (Placebo Comparator): No treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sugammadex — A single dose of sugammadex 2 mg/kg iv
  Other Names: Bridion
  Arms: Sugammadex
Drug: Neostigmine/Glycopyrrolate — A single dose of neostigmine 0.04 mg/kg iv plus glycopyrrolate 0.01 mg/kg iv
  Arms: Neostigmine/glycopyrrolate
Other: Placebo — Placebo
  Arms: No reversal agent

SUMMARY:
Rationale: Recovery from outpatient anesthesia includes dissipation of anesthetics agents, normalization of physiological function, observation for medical or surgical complications, treatment of immediate side effects of anesthesia and surgery and, ultimately, discharge and return home. Street fitness implies that the patient is not only ready to go home, but is also capable of safely taking part in the traffic. A full recovery of cognitive functions is part of this stage. Neuromuscular blocking agents (NMBAs) are commonly used during surgery to facilitate endotracheal intubation, allow assisted or controlled ventilation, and let surgery proceed easily. Sugammadex is approved in Europe for routine clinical use to reverse neuromuscular blockade induced by steroidal non-depolarizing muscle relaxants. Several anesthesiologists from all over the world, have independently reported that patients seem to be more alert in the early phase of recovery after reversal of NMB with sugammadex compared to reversal with a cholinesterase inhibitor or spontaneous recovery. However, these observations have not been substantiated in a clinical study.

Objective: The main aim of the present study is to assess whether sugammadex has a positive effect on the post-operative alertness of the patients, to assess the nature, magnitude and the time of onset of this effect and if a clinically relevant effect has been observed to enable the sample size calculation for a formal well-powered efficacy study.

Study design: Randomized, controlled observer-blind single centre phase IV study. Upon After stratification for type of surgery and age patients will be randomized to receive sugammadex (arm A), neostigmine/glycopyrrolate (Arm B) or no reversal agent (arm C).

Study population: A total of 30 evaluable subjects, aged 18-65 years, with a medical need for general anesthesia and neuromuscular blockade, will be included in the study.

Intervention: Anesthesia will be standardized according to the usual protocol. At the end of the surgery when TOF ratio is ~0,9, and approximately 70-80% of nicotine receptors are still blocked by rocuronium, patients will receive either sugammadex, neostigmine plus glycopyrrolate, or no reversal agent.

Main study parameters: At 30, 60, and 120 minutes after the TOF ratio of ~0,9 has been reached, the following commonly used, and non-invasive cognitive evaluations/scoring lists will be carried out in a subsequent order to assess recovery and psychomotor function: Modified Aldrete Score, the trail making test, the Maddox wing test, and visual analogue scales from both observer and patient.

DETAILED DESCRIPTION:
The number of ambulatory surgical procedures is increasing rapidly. Surgery without one or more overnight stays in hospital is appreciated by most patients and has considerable economic and efficiency advantages. It is facilitated by new anesthetic and analgesic drugs with a more rapid onset and shorter and more reliable duration of action. Paramount for successful ambulatory surgery is the timely discharge of a patient who is at the time of discharge fit to go home.

Early discharge Release of patients, who later experience postoperative complications requiring unanticipated hospital re-admission, should not occur. Fatigue, nausea, vomiting or pain can delay the patient's discharge.2 Patients with psychomotor impairment may be prone to accidents while travelling or at home.3 Short stays are an acceptable practice only if the patient can return home safely and comfortably with minimal side effects from anesthesia and surgery.

Stages of recovery Recovery from outpatient anesthesia includes dissipation of anesthetic agents, normalization of physiological function, observation for medical or surgical complications, treatment of immediate side effects of anesthesia and surgery and, ultimately, discharge and return home.4 Recovery from anesthesia may be divided into three main stages.

Early recovery Awakening and recovery of vital reflexes. Intermediate recovery Intermediate clinical recovery, home readiness. Late recovery Full recovery. Psychological recovery.

Home readiness and street fitness Intermediate recovery implies that the patient is ready to go home (accompanied by a care taker). Street fitness means that the patient is not only ready to go home, but is also capable of safely taking part in the traffic.6 Part of this is full recovery of cognitive functions.

Tests Scoring systems developed to guide the transfer from the hospital recovery room to the ward may be used to assess the early recovery of ambulatory surgical patients. The most commonly used method, described by Aldrete and Kroulik provides objective information on the physical condition of patients arriving in the recovery room after anesthesia.7 This test was modified in 1995 and assigns a score of 0, 1 or 2 to activity, respiration, circulation, consciousness and oxygenation. A score of 9 or 10 indicates adequacy of early recovery and enable discharge from the post-anesthesia care unit (PACU).8 Intermediate recovery to home readiness cannot be determined only with early recovery tests.9 Chung suggested a post-anesthetic discharge scoring system (PADSS), which may provide a reliable measure of anesthetic recovery.10 PADSS is based on vital signs, ambulation and mental status, pain, nausea and vomiting, surgical bleeding and fluid intake and output. The qualifications for discharge include a postoperative discharge score of 9 or more and the presence of a competent adult to accompany the patient home.

Assessment of late recovery (e.g. when the patient is ready to drive a car or resume normal daily activities) requires sophisticated laboratory tests that cannot be used in normal clinical practice.11 Many tests have been applied to assess recovery.

The Human Performance Measurement/Basic Elements of Performance (HPM/BEP) system® (Human Performance Measurement, Inc, Arlington, TX, USA) collects motor performance data. The HPM module for hands (BEP 1) has been used by e.g. Haavisto.12 BEP 1 is a multifunction system designed to measure different aspects of the upper extremity, including visual spatial memory capacity, simple reaction time, choice reaction time, movement speed, wrist tapping and co-ordination. The test-retest reliabilities of HPM/BEP tests were described in detail by Kauranen, and the reliability of the system was acceptable.13 The BEP1 module includes visual spatial memory capacity, simple reaction time, one-choice reaction time 1 speed of movement, two-choice reaction time 1 speed of movement, index finger-tapping speed, co-ordination test, digit-symbol substitution and the Maddox Wing test.

Neuromuscular blocking agents Neuromuscular blocking agents (NMBAs) are commonly used during surgery to facilitate endotracheal intubation, allow assisted or controlled ventilation, and let surgery proceed easily. Although neuromuscular function will recover spontaneously, such recovery is frequently only partial. However, a rapid and complete reversal of neuromuscular blockade (NMB) is desirable in the surgical setting to avoid residual paralysis and related adverse outcomes, amongst them impaired motor behaviour.

Reversal of NMB Traditionally, reversal of NMB has been accomplished with a cholinesterase inhibitor (e.g. neostigmine, pyridostigmine, edrophonium) that acts by inhibiting the breakdown of ACh in the neuromuscular junction.14 Although effective once some recovery has already taken place, cholinesterase inhibitors are associated with a number of limitations, including the induction of cholinergic adverse events (e.g. bradycardia, bronchospasm, bronchial secretions, abdominal cramping) and incomplete reversal of NMB under certain circumstances.15, 16

Sugammadex Sugammadex (Bridion®) has a novel approach to the rapid reversal of steroid based NMBA's.17, 18 The drug has been developed in The Netherlands by Organon, which is now part of Schering-Plough, which is part of Merck. The drug is a modified gamma-cyclodextrin that is water soluble but has a lipophilic cavity that traps the NMBA. The formation of this sugammadex/NMBA complex results in a reduction in the amount of free circulating NMBA, leaving the receptor available for binding to Ach.19 Sugammadex acts selectively against the steroidal NMBAs rocuronium and vecuronium but has little or no activity against nonsteroidal NMBAs (eg, succinylcholine, atracurium, cisatracurium). There is no evidence that sugammadex is metabolized; the drug is primarily eliminated via the renal route as unchanged drug. The drug is in Europe approved for routine clinical use to reverse neuromuscular blockade induced by steroidal non-depolarizing muscle relaxants.

In surgical patients, sugammadex produces dose-dependent reversal of NMB induced by rocuronium or vecuronium.20-22 In comparative studies, sugammadex has demonstrated effectiveness superior to cholinesterase inhibitors for NMB reversal at several time points after the administration of rocuronium or vecuronium. This includes routine reversal of deep or moderate NMB and immediate reversal of NMB.23-25 For example, in the routine reversal of deep NMB, sugammadex was associated with a 15-fold shorter median time to recovery of the T4/T1 ratio to 0.9 compared with neostigmine under sevoflurane anesthesia.

Sugammadex is very well tolerated with no significant cardiovascular or hemodynamic adverse events.26 Dysgeusia (metallic or bitter taste) was the most common adverse event, but this was primarily seen at doses ≥32 mg/kg; there were only a few reports of dysgeusia in surgical patients receiving the drug. Age, gender, race, and ethnicity do not appear to influence the safety of sugammadex.27

Rationale for the study Sugammadex has been registered in The Netherlands since October 2008. Several anesthesiologists from all over the world, have independently reported that patients seem to be more alert in the early phase of recovery after reversal of NMB with sugammadex compared to reversal with a cholinesterase inhibitor or spontaneous recovery. However, these observations have not been substantiated in a clinical study.

It has been proven that at a TOF ratio of 0,9, i.e. when clinical muscle relaxation has nearly disappeared and the patient can be safely extubated, 70-80% of the nicotine receptors are still blocked by the NMBA. An explanation for the possible increase of alertness after reversal with sugammadex could be that sugammadex very efficiently and quickly reverses this rest blockade, resulting in a quick return of alertness and cognitive functions due to an arousal from incoming signals from the γ-motor system. Because sugammadex is inert, it is less likely that an unknown pharmacological effect of sugammadex, a cyclodextrin, is responsible for this supposed effect.

Increased alertness immediately after anesthesia has a positive effect on patient safety and wellbeing and would enable earlier discharge from the PACU. Earlier discharge contributes to an efficient use of the PACU in general and might allow earlier hospital discharge for patients who had surgery in the daycare setting, because they meet the street fitness criteria sooner.

This pilot study has been designed to assess whether sugammadex indeed has, compared with neostigmine or placebo, a positive effect on the street fitness of patients and to assess the nature, magnitude and the time of onset of this effect (if any). 30 patients will be randomized in three groups of 10 patients each (sugammadex, neostigmine/glycopyrrolate and no reversal). These numbers are based on practical considerations, as there are no data available to base a sample size calculation on. The data for this study will enable a sample size calculation for a formal well-powered efficacy study. If a supposed effect on alertness can be demonstrated, it may be worthwhile to investigate the mechanism of action as well.

The investigators have chosen for a trial design in which sugammadex will be used to reverse the neuromuscular blockade induced by rocuronium. Sugammadex in the first, neostigmine/glycopyrrolate in the second, and placebo in the third study arm, will be administered post surgery when clinical neuromuscular function has recovered to the level of TOF ratio ~ 0,9 (i.e. when 70-80% of the receptors are still occupied). It is supposed that sugammadex will efficiently and quickly reverse this "subclinical" rest blockade, leading to an increased alertness. Since a higher alertness has never been described from the traditional drug neostigmine or from placebo is it not expected that they have such an effect. The post surgery cognitive evaluations will be performed 30 minutes after this TOF ratio has been reached. This first 30 minutes time point is considered clinically relevant. In case an effect can only be demonstrated later, the relevance becomes questionable. TOF will only be measured until it reaches approximately 0.9, thereafter only cognitive functions will be evaluated.

A limited number of commonly used cognitive tests have been selected to assess recovery and psychomotor function, including the Modified Aldrete Score, the trail making test, the Maddox wing test and visual analogue scales. With these tests any positive effect of sugammadex on recovery and alertness should be demonstrable.

ELIGIBILITY:
Inclusion Criteria:

* Males and females.
* Age 18-65 years.
* Able to perform the study assessments.
* ASA classification 1 or 2 (Appendix 1).
* Medical need for general anesthesia and neuromuscular blockade.
* NMB with the standard dose of rocuronium. If the surgery lasts longer than 75 minutes the patient will be excluded.
* Minor surgical and gynecological procedures that require tracheal intubation and mechanical ventilation.
* At the pre operative consult the patient will be asked if she is pregnant or if there is a possibility that she is pregnant. If yes, the patient will be excluded.
* Signed informed consent.

Exclusion Criteria:

* Pregnant or lactating women.
* Contra-indications for rocuronium, sugammadex, neostigmine and/or glycopyrrolate.
* Use of toremifene, and/or fusidic acid from 24 hours before till 24 hours after surgery.
* Patients on oral hormonal contraceptives: inability/unwillingness to comply with the instructions for a missed dose according to the SPC text after surgery.
* Patients on non-oral hormonal contraceptives: inability/unwillingness to apply additional non-hormonal contraceptive methods during the 7 days after surgery.
* Concomitant conditions or diseases that might interfere with the study assessments.
* Concomitant treatment with any experimental drug within 4 weeks before surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Street Fitness in surgical patients undergoing general anesthesia after reversal of neuromuscular rest blockade. | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gert J. Scheffer, MD PhD, Principal Investigator — Professor of Anesthesiology, UMC Radboud
Locations (1):
- UMC Sint Radboud, Nijmegen, Gelderland, Netherlands